CLINICAL TRIAL: NCT01916447
Title: A Phase 1, Open-label, Non-randomized, Dose-escalating Safety, Tolerability, and Pharmacokinetic Study of TAS-102 in Combination With CPT-11 and Bevacizumab in Patients With Advanced Gastrointestinal Tumors
Brief Title: A Phase I Study of TAS-102 in Patients With Advanced Gastrointestinal Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPU-TAS-102-109
Record Dates: First submitted 2013-07-19; First posted 2013-08-05 (Estimated); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Gastrointestinal Tumors
Keywords: Angiogenesis Inhibitor; Monoclonal Antibody; Vascular Endothelial Growth Factor A (VEGF-A)
MeSH Terms: interventions — trifluridine tipiracil drug combination; Irinotecan; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAS-102 and CPT-11 with or without Bevacizumab (Experimental)
  Interventions: Drug: TAS-102; Drug: CPT-11; Drug: Bevacizumab

INTERVENTIONS:
Drug: TAS-102 — Escalating doses (20-35 mg/m2/dose, based on tolerability), orally, twice daily on days 1-5 of each 14-day cycle. Number of cycles: until at least one of the discontinuation criteria is met.
Drug: CPT-11 — Escalating doses (30-minute infusion of 120-180 mg/m2/dose, based on tolerability), IV (in the vein) on Day 1 of each 14-day treatment cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Other Names: camptothecin-11, irinotecan
Drug: Bevacizumab — Dose (infusion of 5 mg/kg administered per site standard practice), IV (in the vein) on Day 1 of each 14-day treatment cycle. Number of cycles: until at least one of the discontinuation criteria is met.
  Other Names: Avastin

SUMMARY:
The purpose of this study is to investigate the safety and determine the maximum tolerated dose of TAS-102 administered in combination with CPT-11 in patients with advanced gastrointestinal tumors.

DETAILED DESCRIPTION:
This is an open-label, non-randomized, dose-escalation, Phase 1 study of TAS-102 administered in combination with CPT-11. The study will be conducted in 2 parts: a Dose Escalation Phase (Part 1) to determine the maximum tolerated dose and an Expansion Phase (Part 2) to further evaluate the safety, pharmacokinetics, and preliminary efficacy of the maximum tolerated dose. Patients will be assigned to sequential dose-level cohorts with each cohort corresponding to a pre-specified dose of TAS-102 and CPT-11 combination. Escalation to the subsequent dose level will occur only after the previous dose level is determined to be safe.

ELIGIBILITY:
Inclusion Criteria:

1. Has provided written informed consent
2. Has advanced gastrointestinal tumors refractory to at least 1 chemotherapy
3. ECOG performance status of 0 or 1
4. Is able to take medications orally
5. Has adequate organ function (bone marrow, kidney and liver)
6. Women of childbearing potential must have a negative pregnancy test and must agree to adequate birth control if conception is possible. Males must agree to adequate birth control.

Exclusion Criteria:

1. Has had certain other recent treatment e.g. major surgery, extended field radiation, anticancer therapy, received investigational agent, within the specified time frames prior to study drug administration
2. Presence of serious illnesses or medical condition(s) e.g. brain metastases, systemic infection, heart failure
3. Has unresolved toxicity of greater than or equal to CTCAE Grade 1 attributed to any prior therapies
4. Known sensitivity to TAS-102, CPT-11, Bevacizumab, or their components
5. Is a pregnant or lactating female
6. Has had either partial or total gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose | Through Cycle 1 and Cycle 2 (ie, 4 weeks)
  The maximum tolerated dose is defined as the highest dose level at which less than 33% of the evaluable patients treated experience a dose-limiting toxicity during Cycle 1 or Cycle 2 (ie, during the first 4 weeks) of study drug administration.
Safety monitoring including adverse events, vital signs, and laboratory assessments | Safety is assessed through 30 days following last administration of study medication or until initiation of new anticancer treatment.
  Standard safety monitoring and grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) will be used.

SECONDARY OUTCOMES:
Investigate the safety of TAS-102 and CPT-11 at the MTD administered in combination with Bevacizumab (5 mg/kg IV). | Through 30 days following last administration of study medication or until initiation of new anticancer treatment
  Standard safety monitoring and grading using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) will be used.
Investigate the clinical pharmacokinetics (PK) of TAS-102, CPT-11, and their metabolites. | Blood samples will be collected in Cycle 1 at pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 10, 24 and 48 hours post AM dose of TAS-102 in combination with CPT-11.
  PK analysis for FTD, FTY, TPI, CPT-11, and SN-38 in plasma and will include Cmax, Tmax, AUC0-last, AUC0-inf, and T1/2. FTD and TPI: CL/F, Vd/F will be calculated.
Document any preliminary antitumor activity of TAS-102 administered in combination with CPT-11 and in combination with CPT-11 and Bevacizumab. | After every 4 cycles (i.e., every 8 weeks)
  Tumor assessments using Response Evlauation Criteria in Solid Tumors (RECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Saltz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Los Angeles Clinical Site, Los Angeles, California
  - Chicago Clinical Site, Chicago, Illinois
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee